CLINICAL TRIAL: NCT01548612
Title: Randomised Double Blind Placebo Controlled Study of Sodium Nitroprusside Added to Treatment as Usual in Patients With Schizophrenia
Brief Title: Add-on Sodium Nitroprusside to Treatment as Usual in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jaime Eduardo Cecilio Hallak, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNPSCZ001
Record Dates: First submitted 2012-02-13; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Nitric oxide; Sodium nitroprusside
MeSH Terms: conditions — Schizophrenia | interventions — Nitroprusside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium nitroprusside (Experimental)
  Interventions: Drug: Sodium nitroprusside
- Placebo (Placebo Comparator): Glucose solution 5%
  Interventions: Drug: Glucose solution

INTERVENTIONS:
Drug: Sodium nitroprusside — Intravenous infusion of 0,5 mcg/kg/min for 240 minutes
  Arms: Sodium nitroprusside
Drug: Glucose solution — Intravenous infusion of glucose solution 5% for 240 minutes
  Arms: Placebo

SUMMARY:
In spite of the numerous studies on schizophrenia, its etiology and physiopathology remain unknown. Evidence suggests a possible implication of nitric oxide (NO) in schizophrenia. NO is a gas with unique chemistry and influences the release of neurotransmitters, learning, memory and neurodevelopment. Recent studies that investigated the role of NO in patients with schizophrenia found evidence that points to a disruption in NO-mediated neurotransmission in schizophrenia. Accordingly, we believe that the administration of sodium nitroprusside, an NO donor, will ameliorate schizophrenia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Patients in an acute psychotic episode requiring full hospitalization

Exclusion Criteria:

* Significant medical conditions (heart, kidney, liver, thyroid or neurological diseases, hypovitaminosis B12, hyponatremia)
* Pregnancy
* Breastfeeding
* Previous hypersensitivity to sodium nitroprusside
* DSM-IV diagnosis of drug abuse or dependence

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in BPRS score | baseline and up to 4 weeks
  Brief Psychiatric Rating Scale
Change in PANSS negative subscale score | Every hour for 4 hours, then at +12h, then daily for 7 days, then weekly for 4 weeks
  Positive and Negative Syndrome Scale

SECONDARY OUTCOMES:
Cognitive assessment | Baseline and after 12 h
  FAS, 2-back, Stroop Color Word Test

CONTACTS AND LOCATIONS:
Overall Officials: Jaime EC Hallak, Doctor, Principal Investigator — Ribeirao Preto Medical School, University of Sao Paulo
Locations (1):
- University General Hospital of the Ribeirao Preto Medical School, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Hallak JE, Maia-de-Oliveira JP, Abrao J, Evora PR, Zuardi AW, Crippa JA, Belmonte-de-Abreu P, Baker GB, Dursun SM. Rapid improvement of acute schizophrenia symptoms after intravenous sodium nitroprusside: a randomized, double-blind, placebo-controlled trial. JAMA Psychiatry. 2013 Jul;70(7):668-76. doi: 10.1001/jamapsychiatry.2013.1292. PMID 23699763